CLINICAL TRIAL: NCT00410085
Title: Renal Hemodynamics and Tubular Function in Patients With Obstructive Sleep Apnea and Healthy Controls
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Pia H Gjørup, Department of Medical Research, Holstebro Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MED.RES.HOS.2004.03.PHH
Record Dates: First submitted 2006-12-10; First posted 2006-12-12 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Obstructive Sleep Apnea; Healthy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — omega-N-Methylarginine

INTERVENTIONS:
Drug: L-NMMA (N-mono.methyl-L-arginine)

SUMMARY:
Nitrogen-oxide (NO) plays an important role for blood pressure regulation, renal hemodynamics, and the renal excretion of sodium. NO is synthesized from L-arginine in the vascular endothelium and have a very short half-life in plasma and is therefore very difficult to measure directly.

L-mono-methyl-L-arginine (L-NMMA) is an analogue to L-arginine and a competitive inhibitor of NO, and therefore can be used to study the effect of NO on the circulation. In normal subjects, infusion of L-NMMA will cause an increase in blood pressure, decreased renal plasma-flow, decreased glomerular filtration rate, and a decreased excretion of sodium.

Hypothesis: Patients with obstructive sleep apnea has a decreased activity in the NO-system. This is contributing to the hypertension often seen in these patients. Decreased activity in the NO-system can be revealed by diminished fall in renal hemodynamic and sodium excretion after infusion of L-NMMA.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea

Exclusion Criteria:

* Drug or alcohol abuse
* Pregnancy
* Disease of the heart, lungs, liver, kidney or endocrine organs
* Cerebral infarction
* Diabetes
* Gastrointestinal disease

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-01; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Regional Hospital Holstebro
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Ringkoebing County, Denmark